CLINICAL TRIAL: NCT06304467
Title: Contingency Management for Patients With Alcohol-Associated Liver Disease Following Liver Transplantation
Brief Title: CM for Patients With ALD After Liver Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arpan A. Patel, MD (Other)
Responsible Party: Sponsor-Investigator, Arpan A. Patel, MD, Hepatologist, Assistant Professor, David Geffen School of Medicine at UCLA, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#23-001133
Record Dates: First submitted 2024-02-07; First posted 2024-03-12 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder; Alcohol; Liver; Post Liver Transplant; Contingency Management; Alcohol Liver Disease
Keywords: Alcohol Liver Disease; Contingency Management; Post Liver Transplant; Alcohol Use Disorder; Post Liver Transplant Drinking
MeSH Terms: conditions — Alcoholism; Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment As Usual (TAU) (No Intervention): Study Subjects randomized to treatment as usual (TAU) will not receive an intervention. They will continue with follow-up visits in the outpatient clinic as part of standard of care. .
- Contingency Management (CM) (Experimental): Study subjects who have received a liver transplant and have been randomized to the treatment arm will receive contingency management, a positive reinforcement behavioral treatment with escalating rewards for consecutive either negative urine and blood tests (or lower value of metabolites than the previous week for PeTH) depending on which results are received first, capped at a maximum of $80 (in the form of a gift card) at the week 10 visit.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Study subjects who have received a liver transplant and have been randomized to the treatment arm will receive contingency management, a positive reinforcement behavioral treatment with escalating rewards for consecutive either negative urine and blood tests (or lower value of metabolites than the previous week for PeTH) depending on which results are received first, capped at a maximum of $80 (in the form of a gift card) at the week 10 visit.
  Arms: Contingency Management (CM)

SUMMARY:
Alcohol associated liver disease (ALD) refers to liver injury, such as cirrhosis, that is caused by alcohol use. It affects 2 million adults in the U.S. and is now the leading cause of cirrhosis-related hospitalizations, cirrhosis- related deaths, and liver transplantation. Alcohol use disorder (AUD), the root cause of ALD, affects 15 million Americans each year. While research studies have shown that behavioral therapy and medications specific for alcohol use have helped people overcome their alcohol use disorder, there has not been enough information related to how successful these treatments are specifically for people with ALD. This study will look at a behavioral treatment called "contingency management" (CM) that has shown to be effective with people with other substance use disorders. CM is based on the principles of operant conditioning that involves offering prize-based or monetary incentives to patients with substance use disorders to reduce substance use. This study will look at the efficacy and acceptability of CM in patients who received a liver transplant and have evidence of recurrent alcohol use.

The proposed study is a pilot randomized controlled trial of 30 patients with ALD who received a liver transplant; 15 will be randomized to receive a 10-week CM intervention while 15 will receive treatment as usual (TAU or control). Subjects will be asked to complete 12 study visits (including Screening and Baseline Visits) that will last 1 to 2 hours each depending on the visit. All visits will be completed via Zoom or by phone. Study staff will instruct participants on how to use Zoom, if necessary. During the Screening and Baseline Visits, subjects will be: 1) asked to provide a urine test and blood draw, 2) complete the SCID-5 AUD, a semi-structured interview guide for making the major DSM-5 diagnoses, 3) complete the Iowa Gambling Test which looks at decision-making skills, 4) complete a survey that looks at the subject's quality of life after liver transplant, 4) review how much alcohol the subject has consumed in the last 30 days, 5) and if the subject has received any current AUD treatments. Once the Screening and Baseline visits are completed, subjects will be randomized to either the CM group or the TAU group. During the weekly visits, subjects will be asked to provide blood and urine samples and will be asked if they have had any alcohol since their last visit. All subjects will receive $20 for completing the visits. For those in the CM group, subjects will also receive a CM reward for negative urine and/or blood tests, depending on which results we receive first-with rewards ranging from $5 to $80 depending on the week. Additionally, during weeks 1, 5, and 10, those in the CM group will also complete the Client Satisfaction Questionnaire-8 to assess client satisfaction with CM and complete a semi-structured interview about the CM protocol as well as CM acceptability and feasibility.

DETAILED DESCRIPTION:
This study is a pilot randomized controlled trial of 30 patients with ALD who received a liver transplant; 15 will be randomized to receive a 10-week CM intervention while 15 will receive treatment as usual (control).

Subjects will be recruited directly by research staff as well through MyChart messages.

For in-clinic subjects: Subjects will be identified by the RA via EMR review of patients listed for the day's clinic. Once identified, the Co-Investigator will approach the patient during the outpatient clinic visit with the recruitment flyer. The Co-Investigator will inform the participant that they may be eligible for the study. They will ask patients if the RA may contact them via phone to explain the study in more detail and/or answer any questions the subject may have after reviewing the flyer. If the subject agrees to be contacted, the Co-investigator will notify the RA and let the RA know that the subject has provided consent to contact. The RA will only contact the subject if the Co-Investigator has indicated the subject has provided permission to contact him or her. If the subject has declined permission for contact, the RA will not contact the subject, either by phone or other communication.

Alternatively, the RA may also approach potential subjects identified in clinic. The RA will provide the study flyer, explain the study in detail, and answer any questions the subject may have. If the subject voices interest in participating in the study, the RA can schedule the Consent and Baseline Visit that is mutually agreeable for the subject and RA. The RA will provide study contact information to the subject in case he or she needs to reschedule, or if any issues arise.

Identification by Clinical Staff: The PI will send quarterly emails to the clinical staff of the post-liver transplant clinics which includes physicians, nurse practitioners, social workers, and staff nurses. The email includes a brief summary of the study and the Eligibility Criteria. If the clinical staff have identified any potential subjects, they will email the PI or research assistant who will review the subject's electronic medical record to confirm eligibility. Once screened, the RA will send a MyChart message to the potential subject with study details and study contact information. If the subject is interested in the study and responds to the MyChart message through MyChart, by email, or by phone, then the RA will schedule the Consent and Baseline Visit according to the protocol.

MyChart Messages:

The study team will work with Care Connect analysts to create a work bench report that will identify patients that meet study criteria and the patients on the report will be sent a MyChart Recruitment message. The UCLA Embedded Clinical Research and Innovation (ECRI) team will run the workbench report and send out the messages. Only if the patient replies back with interest will the study team have access to their identifying information to contact them. The research assistant will review the subject's electronic medical record to confirm eligibility. Once screened, the RA will contact the potential subject via MyChart with more details about the study and to ask if they may contact them over the phone to discuss the study and answer any questions they may have. If they respond via MyChart that the RA may contact him or her, the RA will contact them via phone to explain the study, answer any questions, and if the subject is interested, schedule the Consent and Baseline Visit according to the protocol.

After written consent is obtained, the RA will confirm eligibility criteria:

If eligibility is confirmed and signed off by the PI, the participant will complete Baseline Visit activities via Zoom:

1. Record socio-demographic data (self-reported demographics, behavior, and health data) and locator form
2. Complete the Iowa Gambling Task
3. Complete Structured Clinical Interview-5 for AUD (SCID-5 AUD), a semi-structured interview guide for making the major DSM-5 diagnoses
4. Urine sample for EtG
5. Blood draw for PeTH
6. Complete Timeline Followback (TLFB), a validated instrument to assess amounts of drinking within the last 30 days
7. Record concurrent AUD treatment strategies and therapies
8. Complete Patient-Reported Outcomes Measurement Information System (PROMIS), to assess patient's quality of life after liver transplantation. The psychometric properties of this instrument have been previously validated in patients who have received a liver transplant.
9. Randomize participant to contingency management (CM) or treatment as usual (TAU). Participants will be randomly assigned to either the CM treatment group or the TAU group (control) using a SAS® randomization software. Participants will be stratified by applying SCID-5-AUD criteria (groups will be mild or moderate/severe).

All participants will receive a $20 gift card for completing this visit, regardless of treatment arm.

After the initial visit, participants will attend weekly Zoom visits for 10 weeks and will complete assessments according to the protocol. At Visit 2, Visit 5, and Visit 10, participants will also undergo audio recorded semi-structured interviews about the CM protocol as well as CM acceptability and feasibility interviews with the research team. After these interviews, the audio-recordings will be analyzed as part of the study's first aim to look at the acceptability and feasibility of CM in the ALD population.

Since all weekly visits will be completed via Zoom or phone, participants will need to provide blood and urine samples at the nearest UCLA lab before their next weekly visit. CM rewards will not be provided until the study team receives the lab results for that week.

All participants will be compensated for completing each study visit with a gift card regardless of their randomization group. For those in the CM group, participants will also receive a CM reward for negative urine (EtG) and/or blood tests (PeTH), depending on which results are received first. Because PeTH can be elevated for several weeks after a positive test, a lower PeTH value in a subsequent week of checking will be considered a "negative" result, per previous studies. Additionally, if participants in the CM group have negative urine and/or blood test for 2 consecutive weeks, participants will receive a CM bonus.

The primary outcome for the study is the number of non-drinking days, which will be assessed by objective measures (i.e., presence of alcohol biomarkers in the blood and urine), as well as subjective measures (i.e., Timeline Followback). These assessments will be completed weekly. For the 10-week CM intervention, there will be a maximum of 70 non-drinking days.

Secondary outcomes include:

* Health-related quality of life will be assessed using the Patient-Reported Outcomes Measurement Information System at the beginning and end of the intervention,
* Acceptability of the intervention will be assessed with the Client Satisfaction Questionnaire-8 (CSQ-8) with a mean score of 24 (scale: 8-32) which will be considered acceptable, based on prior pilot interventions for AUD, and
* Feasibility of the intervention will be assessed by calculating rates of recruitment and retention throughout the study period.

We will also obtain qualitative descriptions of acceptability and feasibility through individual, semi-structured interviews conducted with all 15 participants in the CM arm during three specific time points (V1, V5, V10).

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older
* Have received a liver transplant
* Has documented return to drinking (subjective or objective) within the past 60 days
* Willing to partake in behavioral treatment for AUD
* Written informed consent and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Current treatment for another substance use disorder
* Unwilling to partake in behavioral treatment for AUD
* Unwilling to provide written informed consent
* Non-English speaking

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Non-Drinking Days | 10 Weeks
  The primary outcome for the study is the number of non-drinking days, which will be assessed by objective measures (i.e., presence of alcohol biomarkers in the blood and urine), as well as subjective measures (i.e., Timeline Followback). For the 10-week CM intervention, there will be a maximum of 70 non-drinking days.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS® 29+2 Profile v2.1 (PROPr)) | 10 Weeks
  To assess health related quality of life. The PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain.
Client Satisfaction Questionnaire-8. | 10 Weeks
  To assess acceptability of the CM program. An overall score is calculated by summing the respondent's rating (item rating) score for each scale item. For the CSQ-8 version, scores therefore range from 8 to 32, with higher values indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Arpan G Patel, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Pfleger Liver Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No